CLINICAL TRIAL: NCT00254644
Title: Morphofunctional Imaging and Developmental Dyslexia
Acronym: PHR04-CH/DYS
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: PHRR04-CH/DYS
Record Dates: First submitted 2005-11-15; First posted 2005-11-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2011-05

CONDITIONS: Developmental Dyslexia
Keywords: phonological treatment; language; fMRI
MeSH Terms: conditions — Dyslexia; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dyslexia: adults from 18-35 ans.
  Interventions: Procedure: Morphological and functional MRI
- Control: adults from 18-35 ans.
  Interventions: Procedure: Morphological and functional MRI

INTERVENTIONS:
Procedure: Morphological and functional MRI — one time

SUMMARY:
Developmental dyslexia is a frequent learning disability. The aim of this study is to analyze cortical thickness and phonological treatment in right handed adults with developmental dyslexia. They are compared to control adults paired with age and laterality. To study phonological treatment, the researchers used functional magnetic resonance imaging (fMRI) with a rime judgement task and silent word generation.

ELIGIBILITY:
Inclusion Criteria:

* Developmental dyslexia according to Critchley.
* Normal performance intelligence quotient (PIQ)
* Age: 18-35 years
* Sex: Male
* Right handed
* No hearing deficit.

Exclusion Criteria:

* No head injury
* No attention deficit hyperactivity disorder (ADHD)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a prospective study including 15 right-handed male subjects, aged 18 to 35 years, carrying a developmental dyslexia and 15 control subjects handed the same sex. We chose to include only male subjects to obtain a homogeneous population and to avoid the problem of a functional organization differs according to gender.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Cortical thickness | 2 years
  The average cortical thickness maps of healthy subjects and dyslexic will be compared hemisphere by hemisphere. This will identify whether there are cortical areas including cortical thickness differed significantly between normal and dyslexic.ts of different ages

SECONDARY OUTCOMES:
Average cortical thickness | 2 years
  For each group, cortical thickness maps of average left and right hemispheres are compared. This will identify whether there is an asymmetry left / right in terms of cortical thickness in normal subjects and dyslexic.

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Bonnet-Brilhault, Principal Investigator — CHU Tours
Locations (1):
- CHU, Tours, France